CLINICAL TRIAL: NCT01260662
Title: Randomized Blinded Three Arm Trial of Propofol, 1:1 Combination of Propofol and Ketamine, and 4:1 Combination of Propofol and Ketamine for Procedural Sedation in the Emergency Department
Brief Title: Randomized Clinical Trial of Propofol, 1:1 and 4:1 Combination of Propofol and Ketamine for Procedural Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR 10-3230
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Procedural Sedation
Keywords: Deep Procedural Sedation; Propofol; Ketamine; Emergency Department; Monitoring; Capnography; Procedural Sedation in the Emergency Department
MeSH Terms: conditions — Emergencies | interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol (Active Comparator): Deep sedation using propofol
  Interventions: Drug: Propofol
- 1:1 Propofol/Ketamine (Experimental): Propofol and ketamine mixed 1:1, given at 0.1 cc/kg as initial bolus, followed by 1/2 that dose every 3 minutes as need for sedation
  Interventions: Drug: 1:1 Propofol/Ketamine
- 4:1 Propofol/Ketamine (Experimental): Propofol and ketamine mixed 4:1, given at 0.1 cc/kg as initial bolus, followed by 1/2 that dose every 3 minutes as need for sedation
  Interventions: Drug: 4:1 Propofol/Ketamine

INTERVENTIONS:
Drug: Propofol — 1 mg/kg IV bolus followed by 0.5 mg/kg every 3 minutes as need for sedation
  Arms: Propofol
Drug: 1:1 Propofol/Ketamine — Propofol and ketamine mixed 1:1, given at 1 mg/kg IV bolus followed by 0.5 mg/kg every 3 minutes as need for sedation
  Arms: 1:1 Propofol/Ketamine
Drug: 4:1 Propofol/Ketamine — Propofol and ketamine mixed 4:1, given at 1 mg/kg IV bolus followed by 0.5 mg/kg every 3 minutes as need for sedation
  Arms: 4:1 Propofol/Ketamine

SUMMARY:
This will be a randomized trial of propofol versus the combination of propofol and ketamine for procedural sedation for procedures in the Emergency Department (ED). Propofol produces sedation, hypnosis, and dense amnesia, and is commonly used in the ED at Hennepin County Medical Center (HCMC) for procedural sedation. Ketamine is a dissociative anesthetic that is also frequently used in the ED in children and sometimes in adults. It has been proposed that by combining the two agents, the negative side effects of respiratory depression and hypotension associated with propofol, and the negative effects of dysphoria and vomiting associated with ketamine, can be avoided.

In the proposed study, patients seen in the ED who will require procedural sedation for a painful procedure will be randomized to receive either propofol or propofol and ketamine. During the procedure, patients will be monitored per the standard of care, including use of a cardiac monitor, non-invasive blood pressure monitoring, pulse oximetry, nasal sample end-tidal carbon dioxide, and physician assessment. Once the procedure is successfully completed and the patient has returned to his/her baseline mental status, the patient will be asked to mark a 100 mm visual analog scale regarding perceived pain during the procedure, memory of the procedure, and overall satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing procedural sedation for an urgent procedure in the Emergency Department

Exclusion Criteria:

* Allergy to propofol or ketamine, intoxication, altered mental status, ASA physical status score >2

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miner JR, Moore JC, Austad EJ, Plummer D, Hubbard L, Gray RO. Randomized, double-blinded, clinical trial of propofol, 1:1 propofol/ketamine, and 4:1 propofol/ketamine for deep procedural sedation in the emergency department. Ann Emerg Med. 2015 May;65(5):479-488.e2. doi: 10.1016/j.annemergmed.2014.08.046. Epub 2014 Oct 16. PMID 25441247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 300 patients recruited in the Emergency Department from October 24, 2010 to February 4, 2013
Pre-assignment Details: 271 enrolled subjects underwent procedural sedation
Groups:
- Propofol: Deep sedation using propofol (10 mg /mL)
  Subjects received a 1 mg/kg IV bolus of propofol followed by 0.5 mg/kg every 3 to 5 minutes as needed to achieve and maintain adequate sedation
- 1:1 Propofol/Ketamine: Deep sedation using 1:1 propofol to ketamine mixture (prepared with propofol 10 mg/mL and ketamine 10mg/mL)
  Subjects received a 1 mg/kg IV bolus of 1:1 propofol/ketamine mixture followed by 0.5 mg/kg every 3 to 5 minutes as needed to achieve and maintain adequate sedation
- 4:1 Propofol/Ketamine: Deep sedation using 4:1 propofol to ketamine mixture (prepared with propofol 10 mg/mL and ketamine 10mg/mL)
  Subjects received a 1 mg/kg IV bolus of 4:1 propofol/ketamine mixture followed by 0.5 mg/kg every 3 to 5 minutes as needed to achieve and maintain adequate sedation
Period: Overall Study
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Started | 90 | 85 | 96
Completed | 90 | 85 | 96
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Participants include any individual who received drug and underwent procedural sedation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine | Total
Number analyzed (Participants) | 90 | 85 | 96 | 271
Age, Continuous [Mean (Full Range); unit: years] | 40 [18 to 83] | 39 [18 to 80] | 36 [18 to 84] | 38 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 45 | 128
  Male | 47 | 45 | 51 | 143
Region of Enrollment [Number; unit: participants]
  United States | 90 | 85 | 96 | 271

OUTCOME MEASURES:

1. Primary Outcome: Clinical Interventions During Sedation
Description: Add/increase in supplemental oxygen, stimulation to induce respiration, airway repositioning, assisted ventilations, endotracheal intubation
Time Frame: From start of sedation procedure to end of sedation procedure, up to 24 hours
Population: 100 subjects were randomized to each group, 90 subjects in the propofol arm completed the study, 85 in the 1:1 propofol/ketamine arm, and 96 in the 4:1 propofol/ketamine arm
Measure: Number; unit: Clinical interventions performed
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Number analyzed (Participants) | 90 | 85 | 96
Clinical interventions performed | 41 | 33 | 48

2. Primary Outcome: Hypoxia
Description: Pulse oximetry
Time Frame: From start of sedation procedure to end of sedation procedure, up to 24 hours
Population: as for outcome 1
Measure: Number; unit: Patients which experienced hypoxia
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Number analyzed (Participants) | 90 | 85 | 96
Patients which experienced hypoxia | 11 | 6 | 18

3. Secondary Outcome: Respiratory Depression
Description: Continuous capnographic monitoring
Time Frame: From start of sedation procedure to end of sedation procedure, up to 24 hours
Population: as for outcome 1
Measure: Number; unit: number of respiratory depression events
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Number analyzed (Participants) | 90 | 85 | 96
number of respiratory depression events | 15 | 16 | 21

4. Secondary Outcome: Procedural Recall
Description: After patients returned to baseline mental status they were asked whether they were able to recall any of the procedure. Question was answered in a yes or no format.
Time Frame: Immediately after the end of the procedure, a single time point within 30 minutes of procedures conclusion.
Population: as for outcome 1
Measure: Number; unit: percentage report recall of procedure
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Number analyzed (Participants) | 90 | 85 | 96
percentage report recall of procedure | 6 | 14 | 11

ADVERSE EVENTS:
Arm/Group | Propofol | 1:1 Propofol/Ketamine | 4:1 Propofol/Ketamine
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/85 | 0/96
Other Adverse Events (participants affected / at risk) | 0/90 | 0/85 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No